CLINICAL TRIAL: NCT01885351
Title: An Interactive Preventive Health Record to Increase Colorectal Cancer Screening
Acronym: MyCRCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HM14658; R01CA166375-01A1 (NIH); MYCRCS-302259 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2013-04-23; First posted 2013-06-24 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal Cancer Screening; Ambulatory Care; Patient-Centered Care; Intervention Studies; Longitudinal Studies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase II: MyCRCS+Prefs (Experimental): Patients who are identified by the IPHR as study participants will see an attractive link. In the Prefs arm, via question prompt lists, patients will first identify their CRCS preference using previously developed elicitation strategies.
  Tailoring will be used to increase salience of information, motivation, communication, and action plans. We envision the Prefs+ arm in its entirety will be 5-7 minutes, but will depend on Phase I formative work. If the patient remains non-adherent, they will receive an e-mail reminder generated by the IPHR (specific text and frequency determined in Phase I). The Prefs content is identical to the preference portion of the Prefs+Barriers arm, which will allow us to assess the incremental benefit of addressing preferences only and the incremental benefit of addressing preferences and barriers.
  Interventions: Behavioral: MyCRCS+Prefs
- Phase II: MyCRCS+Prefs+Barriers (Experimental): Patients who are identified by the IPHR as study participants will see an attractive link. In the Prefs+Barriers arm, via question prompt lists, patients will first identify their CRCS preference using previously developed elicitation strategies, and subsequently based on their test preference determine their top 3 test-specific barriers/concerns in "real time".
  Tailoring will be used to increase salience of information, motivation, communication, and action plans. We envision the Prefs+Barriers arm in its entirety will be 15-25 minutes, but will depend on Phase I formative work. If the patient remains non-adherent, they will receive an e-mail reminder generated by the IPHR (specific text and frequency determined in Phase I). The Prefs content is identical to the preference portion of the Prefs+Barriers arm, which will allow us to assess the incremental benefit of addressing preferences only and the incremental benefit of addressing preferences and barriers
  Interventions: Behavioral: MyCRCS+Prefs+Barriers
- Phase II: Usual Care (No Intervention): The IPHR will be programmed so that where the IPHR-CRCS would normally present patients, who based on their demographics and health conditions, with content advising them to seek CRCS and links to third-party sites, they would instead be randomized to receive the usual care (IPHR-CRCS).

INTERVENTIONS:
Behavioral: MyCRCS+Prefs — Patients who are identified by the IPHR as study participants will see an attractive link. In the Prefs arm, via question prompt lists, patients will first identify their CRCS preference using previously developed elicitation strategies.
  Tailoring will be used to increase salience of information, motivation, communication, and action plans. We envision the Prefs+ arm in its entirety will be 5-7 minutes, but will depend on Phase I formative work. If the patient remains non-adherent, they will receive an e-mail reminder generated by the IPHR (specific text and frequency determined in Phase I). The Prefs content is identical to the preference portion of the Prefs+Barriers arm, which will allow us to assess the incremental benefit of addressing preferences only and the incremental benefit of addressing preferences and barriers.
  Arms: Phase II: MyCRCS+Prefs
Behavioral: MyCRCS+Prefs+Barriers — Patients who are identified by the IPHR as study participants will see an attractive link. In the Prefs+Barriers arm, via question prompt lists, patients will first identify their CRCS preference using previously developed elicitation strategies, and subsequently based on their test preference determine their top 3-5 test-specific barriers/concerns in "real time".
  Tailoring will be used to increase salience of information, motivation, communication, and action plans. We envision the Prefs+Barriers arm in its entirety will be 15-25 minutes, but will depend on Phase I formative work. If the patient remains non-adherent, they will receive an e-mail reminder generated by the IPHR (specific text and frequency determined in Phase I). The Prefs content is identical to the preference portion of the Prefs+Barriers arm, which will allow us to assess the incremental benefit of addressing preferences only and the incremental benefit of addressing preferences and barriers.
  Arms: Phase II: MyCRCS+Prefs+Barriers

SUMMARY:
This study involves 3 phases that modifies current Interactive Preventative Health Record-Colorectal Cancer Screening (IPHR-CRCS) modules to address each patient's individual colorectal cancer screening (CRCS) knowledge, attitudes, preferences, and test-specific barriers. The study will engage patients, ages 50-75 years who are non-adherent to CRCS, to assess their CRCS test preferences and corresponding test-specific barriers in "real time". Based on patient characteristics (e.g. age, personal and family history, physician CRCS recommendation, CRCS test preferences, top test-specific barriers), tailored messages/videos will appear in the pop-up screens to address/reduce the top patient-reported, test-specific CRCS barriers while incorporating an action plan for CRCS adherence. The investigators hypothesize that modifying the IPHR-CRCS module to address each patient's individual CRCS knowledge, attitudes, preferences, and test-specific barriers will further increase CRCS.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50-75 years
* Non-adherent to CRCS guidelines (i.e., no FOBT in last year, no sigmoidoscopy or barium enema in last 5 years, and no colonoscopy in last 10 years)
* English-speaking
* Have computer access (e.g. home, work, library)
* Additional eligibility for Phase I: focus group participants will be ineligible for the subsequent prototype testing and cognitive/usability testing interviews
* Additional eligibility for Phase I: prototype testing participants will be ineligible for the cognitive/usability testing interviews
* Additional eligibility for Phase II: Seen in the clinic in the last 2 years

Exclusion Criteria:

* Personal CRC history
* Additional exclusion for Phase III: Patients seen at any clinic participating in Phase II

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
CRCS adherence provided by the electronic medical record | Phase II: Baseline up to 12 months post randomization
  Having had ≥1 test (i.e., fecal occult blood test, sigmoidoscopy, colonoscopy and barium enema) within the time frame specified for each procedure will count as adherent CRCS.
CRCS adherence provided by the electronic medical record | Phase III: Baseline up to 12 months post intervention
  Having had ≥1 test (i.e., fecal occult blood test, sigmoidoscopy, colonoscopy and barium enema) within the time frame specified for each procedure will count as adherent CRCS.

SECONDARY OUTCOMES:
Self-reported CRCS adherence | Phase II: Baseline, 3 months, and 9 months post randomization
  The four NCI-recommended CRCS history questions will be included on the self-report surveys. Respondents will identify the last time they had each test (i.e., fecal occult blood test, sigmoidoscopy, colonoscopy and barium enema). Having had ≥1 test within the time frame specified for each procedure will count as adherent CRCS.
EHR Paradata | Phase II: continuous
  We will track participants' use of the intervention and usual care arms to capture number of log-ins, pages viewed, length of view, links clicked. In addition to elucidating patients' uptake of intervention components, these data can indicate engagement for dose-response analyses or be examined as potential mediators. For Phase II, this data will allow us to assess the timing of intervention reminders to make a decision about what frequency is most appropriate so that we can modify before we begin the feasibility study (phase III).
Psychosocial Constructs | Phase II: Baseline, 3 months, and 9 months post randomization
  Scales (e.g. Decisional conflict, intentions , self-efficacy, perceived susceptibility, worry, etc.) are included in the patient questionnaire, which have good psychometric properties.
General and test-specific colorectal cancer screening barriers | Phase II: Baseline, 3 months, and 9 months post randomization
  A previously validated modality-specific colorectal cancer screening barrier instrument will be used. The FOBT-specific scale includes 19 questions relating to barriers for fecal occult blood test, and the colonoscopy-specific scale includes 21 questions relating barriers to colonoscopy. All items are measured on a 5-point Likert-type scale, with 5 representing greater barrier endorsement. Items are summated to create continuous scale scores (range: FOBT=19-95; colonoscopy=21-105).
Self-reported CRCS adherence | Phase III: Baseline and 9 months post intervention
  The four NCI-recommended CRCS history questions will be included on the self-report surveys. Respondents will identify the last time they had each test (i.e., fecal occult blood test, sigmoidoscopy, colonoscopy and barium enema). Having had ≥1 test within the time frame specified for each procedure will count as adherent CRCS.
EHR Paradata | Phase III: Continuous
  We will track participants' use of the intervention and usual care arms to capture number of log-ins, pages viewed, length of view, links clicked. In addition to elucidating patients' uptake of intervention components, these data can indicate engagement for dose-response analyses or be examined as potential mediators. For Phase II, this data will allow us to assess the timing of intervention reminders to make a decision about what frequency is most appropriate so that we can modify before we begin the feasibility study (phase III).
Psychosocial Constructs | Phase III: Baseline and 9 months post intervention
  Scales (e.g. Decisional conflict, intentions , self-efficacy, perceived susceptibility, worry, etc.) are included in the patient questionnaire, which have good psychometric properties.
General and test-specific colorectal cancer screening barriers | Phase III: Baseline and 9 months post intervention
  A previously validated modality-specific colorectal cancer screening barrier instrument will be used. The FOBT-specific scale includes 19 questions relating to barriers for fecal occult blood test, and the colonoscopy-specific scale includes 21 questions relating barriers to colonoscopy. All items are measured on a 5-point Likert-type scale, with 5 representing greater barrier endorsement. Items are summated to create continuous scale scores (range: FOBT=19-95; colonoscopy=21-105).
Feasibility of MyCRCS+ in target setting - patient survey | Phase III: Baseline and 9 months post intervention
  Phase III is a feasibility study to determine among other things, implementation in the "real world" setting. The outcomes we propose to measure are defined by the RE-AIM model. Specifically, we selected four essential elements pertaining to the feasibility of fielding MyCRCS+: Reach, Effectiveness, Implementation, and Maintenance.
  The patient survey will include key questions related to intervention reach and potential future implementation adaptations addressing patient awareness and perception of the practices' MyCRCS+ integration strategies.Surveys will assess: patients' awareness of MyCRCS+, how they learned about it, what they liked or disliked about how practices promoted and used MyCRCS+; to what extent they used the MyCRCS+, the factors that influenced use, facilitators and barriers to both using and acting on MyCRCS+ recommendations; anxiety and worry; and quality of life (QOL).

OTHER OUTCOMES:
Development of MyCRCS+ intervention content | Phase I (months 1-17)
  Develop and pretest MyCRCS+, which focuses on integrating patient CRCS preferences and test-specific barriers in an interactive web-based intervention. Answer the question: What intervention content and reminder content, packaging and frequency are acceptable to patients?

CONTACTS AND LOCATIONS:
Overall Officials: Resa M Jones, MPH, PhD, Principal Investigator — Temple University and Virginia Commonwealth University
Locations (2):
- United States (2):
  - Temple University - General Internal Medicine, Philadelphia, Pennsylvania
  - Virginia Ambulatory Care Outcomes Research Network, Richmond, Virginia